CLINICAL TRIAL: NCT00324142
Title: A Pilot Study of Oral Tinidazole for Women With Recurrent Bacterial Vaginosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Terminated Prematurely
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN-06JGunt-01-B
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Recurrent Bacterial Vaginosis
Keywords: Bacterial vaginosis; Tinidazole; Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis | interventions — Tinidazole

INTERVENTIONS:
Drug: Oral tinidazole

SUMMARY:
This is a study of the drug tinidazole for women with recurrent bacterial vaginosis. Half of the participants will get the drug for 10 days, the other half will get the drug for 10 days and then twice a week for 12 weeks.

DETAILED DESCRIPTION:
This study will recruit 60 women with recurrent bacterial vaginosis. These women must have a current infection to be enrolled in the study and have had two other infections within the past 12 months. After initial screening to make sure that the vaginal symptoms are due to bacterial vaginosis and not the results of a different infection, all of the women will receive tinidazole (a drug that is similar to metronidazole) by mouth for 10 days. At the end of the 10 days, patients will be re-examined. Those women who are free of bacterial vaginosis will enter the second phase of the study, where half of the patients will continue to take tinidazole twice a week for twelve weeks and the other half will take no medication. During this time participants will be examined by the study doctor every 4 weeks to see how effective the treatment has been at preventing the recurrence of bacterial vaginosis. At the end of the 12 weeks, women who are still free of bacterial vaginosis will be seen for 3 more visits over 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Current infection with bacterial vaginosis
* 2 previous episodes of bacterial vaginosis within the past 12 months
* Willing to use contraception
* Able to swallow pills
* Willing to refrain from douching or using vaginal products
* Willing to refrain from alcohol consumption 24 hours before and for 72 hours after taking study medication (tinidazole)

Exclusion Criteria:

* Women with same sex partners
* Menstruating at initial exam
* Presence of yeast, a sexually transmitted disease, or other vaginal infection
* Purulent cervical discharge
* Use of any drug for bacterial vaginosis or yeast within the past 2 weeks prior to enrollment
* Pregnant or nursing
* Taking lithium
* Taking blood thinners (anticoagulation therapy)
* Use of any investigational drug within the previous 30 days
* Active HPV infection requiring treatment
* Use of drugs that suppress the immune system
* History of alcoholism
* Taking disulfiram

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Efficacy of oral tinidazole for treatment of recurrent bacterial vaginosis
Efficacy of oral tinidazole for prevention of recurrent bacterial vaginosis

SECONDARY OUTCOMES:
Patient satisfaction with tinidazole for recurrent bacterial vaginosis

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gunter, MD, Principal Investigator — Kaiser Permamente
Locations (1):
- Kaiser Permanente, San Francisco, California, United States